CLINICAL TRIAL: NCT00208624
Title: Rhythm Disturbances After Ventricular Septal Defects
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kevin O. Maher, MD, Principal Investigator, Emory University
Other Study IDs: 04-118
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Heart Block After Surgery
Keywords: arrhythmia; pediatrics; cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
We would like to conduct a retrospective chart review examining the incidence of surgical heart block in children treated in the Cardiac Service Line at Children's Healthcare of Atlanta. We would like to look at the last 30 surgical heart block cases seen at Children's Healthcare of Atlanta. We will collect the following information on each patient:

Patient Date of Birth Date of the surgical procedure

Weight of the patient at the time of surgery Concomitant Diagnoses Need for permanent pacemaker Outcome of pacing (i.e. pacing successful)

We hope to look at each data element in order to determine potential risks factors for surgical heart block. By identifying the risk factors, the investigator hopes to establish a training program regarding surgical avoidance of certain areas of the heart (if possible) and education regarding pacemaker follow-up.

Each patient will be given a unique study number. The patient's name, social security number, medical record number or initials will not be used in our research database.

ELIGIBILITY:
Inclusion Criteria:

Patients with heart block after surgery -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-12; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maher, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States